CLINICAL TRIAL: NCT01902797
Title: Malaria Survey in the Tak Province Refugee Camps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMRU 1303
Record Dates: First submitted 2013-07-10; First posted 2013-07-18 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Malaria
Keywords: Refugee camps; Household residence; Treated bednets; PCR
MeSH Terms: conditions — Malaria | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Household (Experimental): In each camp, the camp residences are divided into different sections (as clusters for sampling) by camp registration. In the first stage, sections are selected using Population-proportion-to size (PPS) method. In the second stage, households are randomly selected from the household list in each section provided by NGO and local committee. When a household is not responding, a nearest household on the north will be used as replacement. All family members and overnight guests aged above 5 years in the selected household will be invited for venous blood sample (2 ml); for children aged 1-5 years old, the blood sample (100 microL) will be obtained by finger prick; children younger than 1 year old are excluded. The head of household will be invited for a short questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants will be invited to complete questionnaires and those who are over 5 year of age will be asked to give blood samples.

SUMMARY:
According to the World Malaria Report, there were significant decreases in the number of P.falciparum (PF) malaria cases worldwide in the past decade. On the Thai-Myanmar border where transmission is low and seasonal and where incidence of Multi-drugs resistant P.falciparum parasites is the highest, the same trend has been observed with a clear decline in malaria episodes and the ratio of P. falciparum/P. vivax (PF/PV.

Economic development, unprecedented financial support, renewed efforts in vector control, a wider use of rapid diagnosic tests (RDTs) for malaria and the deployment of artemisinin based combination treatments (ACT) are the main contributing factors to those successes against malaria.

However the emergence in Cambodia and on the Thai-Myanmar border of P.falciparum isolates that exhibit resistance to artesunate is threatening those gains . This is characterized by a slow parasite clearance rate observed in patients treated with artesunate.

At the same time, recent SMRU surveys along the Thai-Burmese border using a new cutting-edge technology i.e. highly sensitive quantitative Real Time PCR (RT-PCR) able to detect very low parasitaemia (10 parasites per ml), found up to a 3-5 fold increase in the prevalence of malaria compared to what is found with the usual diagnostic tools such as microscopy, RDT or even conventional PCR.

It seems that a large number of asymptomatic carriers with very low parasites counts (a large potential malaria reservoir) go undetected. If confirmed, this might pose the greatest obstacle for malaria elimination in the region and containment of artemisinin resistance.

The purpose of the survey is to further study and understand the epidemiology of malaria in the refugee camp population using cutting-edge technology (RT-PCR) .

DETAILED DESCRIPTION:
According to the World Malaria Report, there were significant decreases in the number of P.falciparum (PF) malaria cases worldwide in the past decade. On the Thai-Myanmar border where transmission is low and seasonal and where incidence of Multi-drugs resistant P.falciparum parasites is the highest, the same trend has been observed with a clear decline in malaria episodes and the ratio of P. falciparum/P. vivax (PF/PV).

Economic development, unprecedented financial support, renewed efforts in vector control, a wider use of rapid diagnosic tests (RDTs) for malaria and the deployment of artemisinin based combination treatments (ACT) are the main contributing factors to those successes against malaria.

However the emergence in Cambodia and on the Thai-Myanmar border of P.falciparum isolates that exhibit resistance to artesunate is threatening those gains . This is characterized by a slow parasite clearance rate observed in patients treated with artesunate.

At the same time, recent SMRU surveys along the Thai-Burmese border using a new cutting-edge technology i.e. highly sensitive quantitative Real Time PCR (RT-PCR) able to detect very low parasitaemia (10 parasites per ml), found up to a 3-5 fold increase in the prevalence of malaria compared to what is found with the usual diagnostic tools such as microscopy, RDT or even conventional PCR.

It seems that a large number of asymptomatic carriers with very low parasites counts (a large potential malaria reservoir) go undetected. If confirmed, this might pose the greatest obstacle for malaria elimination in the region and containment of artemisinin resistance.

The purpose of the survey is to further study and understand the epidemiology of malaria in the refugee camp population using cutting-edge technology (RT-PCR) .

The necessity of research in Humans With the double mission of malaria elimination and artemisinin-resistance containment, there are intensive malaria activities currently implemented in the refugee camps in the Tak province (a province in Thailand that is on the Thai-Burmese border). The malaria risk among the refugee camp is higher than the Thai residences inside Thailand.

To avoid resource wastage, it is thus essential to conduct a simple questionnaire to understand the current situation of malaria prevention in the camps, especially information regarding the mosquito net ownership and usage (mosquito net distribution has been a major malaria prevention activity among the NGOs in the camps).

PCR method is being used more and more in recent year due to its sensitivity compared to slide reading. PCR is considered being able to capture more cases with sub-microscopic infection. However, the current PCR methods conventionally used in malaria survey usually use finger prick to obtain only few microliters of capillary blood , the detectable level of parasitaemia is therefore limited due to minimal amount of blood from which Plasmodium DNA can be extracted. Thus the RT-PCR method proposed here using 2ml venous blood well compensates these shortcomings.

The comparison of test results of conventional microscopy (currently still as the universal golden standard in the clinics) and RT-PCR will not only enable detection of both symptomatic and asymptomatic malaria cases but help define the epidemiology apart from our conventional understanding of malaria.

Thus this study is necessary and is strategically important for the next roadmap development of malaria elimination and resistance containment.

ELIGIBILITY:
Inclusion Criteria:

* Head of household and all family members
* Overnight guests
* Age > 12 months
* Willing to participate in the study and sign informed consent

Exclusion Criteria:

* All children < 1 year
* Anyone reported history of abnormal blood coagulation
* Anyone who does not consent to participate in the survey

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 908 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Malaria prevalence | 1 day
  Comparison of malaria prevalence by conventional microscopy and RT-PCR to determine the malaria epidemiology in the population

SECONDARY OUTCOMES:
Determine the percentage of households with at least one long lasting insecticide treated nets (LLIN) or insecticide treated nets (ITNs | 1 day
  • percentage of households with at least one long lasting insecticide treated nets (LLIN) or insecticide treated nets (ITNs) per 2 persons
Determine the percentage of refugees sleeping under an ITN/LLIN previous night | 1 day
  Percentage of refugees sleeping under an ITN/LLIN previous night
Determine the percentage of refugees who can recall at least 1 key messages on malaria control and containment/elimination | 1 day
  The percentage of refugees who can recall at least 1 key messages on malaria control and containment/elimination
Determine percentage of refugees who stay overnight outside the camp | 1 day
  The percentage of refugees who stay overnight outside the camp

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Proux, PhD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Refugee Camps, Mae Sot, Changwat Tak, Thailand